CLINICAL TRIAL: NCT02899988
Title: A Phase 2, Multicenter, Randomized, Parallel-Arm, Placebo- Controlled Study of LY3074828 in Subjects With Moderate-to- Severe Plaque Psoriasis
Brief Title: A Study of Mirikizumab (LY3074828) in Participants With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16481; I6T-MC-AMAF (Other: Eli Lilly and Company); 2016-001098-34 (EudraCT Number)
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Results first posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2019-08-15

CONDITIONS: Plaque Psoriasis
Keywords: IL-23; dermatology
MeSH Terms: interventions — mirikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 30 mg Mirikizumab (Experimental): 30 mg Mirikizumab administered subcutaneously (SC) every 8 weeks (Q8W).
  Interventions: Drug: Mirikizumab
- 100 mg Mirikizumab (Experimental): 100 mg Mirikizumab administered SC Q8W.
  Interventions: Drug: Mirikizumab
- 300 mg Mirikizumab (Experimental): 300 mg Mirikizumab administered SC Q8W.
  Interventions: Drug: Mirikizumab
- Placebo (Placebo Comparator): Placebo administered SC Q8W.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirikizumab — Administered SC
  Other Names: LY3074828
  Arms: 100 mg Mirikizumab; 30 mg Mirikizumab; 300 mg Mirikizumab
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy of the study drug mirikizumab in participants with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Present with chronic plaque psoriasis based on an investigator confirmed diagnosis of chronic psoriasis vulgaris for at least 6 months prior to baseline and meet the following criteria:

  * plaque psoriasis involving ≥10% body surface area (BSA) and absolute PASI score ≥12 in affected skin at screening and baseline
  * sPGA score of ≥3 at screening and baseline
* Candidate for biologic treatment for psoriasis.

Exclusion Criteria:

* Have a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute a risk when taking investigational product or could interfere with the interpretation of data.
* Breastfeeding or nursing (lactating) women.
* Have had serious, opportunistic, or chronic/recurring infection within 6 months prior to screening.
* Have received live vaccine(s) (included attenuated live vaccines) within 1 month of screening or intend to during the study.
* Have any other skin conditions (excluding psoriasis) that would affect interpretation of the results.
* Have received systemic nonbiologic psoriasis therapy or phototherapy within 28 days prior to baseline.
* Have received topical psoriasis treatment within 14 days prior to baseline.
* Have received anti-tumor necrosis factor (TNF) biologics, or anti-interleukin (IL)-17 targeting biologics within 8 weeks prior to baseline.
* Have previous exposure to any biologic therapy targeting IL-23 (including ustekinumab), either licensed or investigational (previous briakinumab use is permitted).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2019-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (37):
- United States (12):
  - Renstar Medical Research, Ocala, Florida
  - Forward Clinical Trials, Inc, Tampa, Florida
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - The South Bend Clinic, South Bend, Indiana
  - DS Research, Louisville, Kentucky
  - Dr. Shondra Smith MD, Lake Charles, Louisiana
  - Central Dermatology PC, St Louis, Missouri
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Clinical Partners LLC, Johnston, Rhode Island
  - Menter Dermatology Research Institute, Dallas, Texas
  - Dermatology Associates, Seattle, Washington
- Canada (6):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Calgary
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Halifax
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Montreal
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Peterborough
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Richmond Hill
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Waterloo
- Germany (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt am Main
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mahlow
- Japan (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gifu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kurume
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morioka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagoya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shinagawa-KU
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shinjuku-ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Takaoka-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tsu
- Poland (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Świdnik
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- Puerto Rico (2):
  - Grupo Dermatologico de Carolina, Carolina
  - Ponce School of Medicine CAIMED Center, Ponce

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction: Placebo: Induction: Participants received placebo subcutaneously (SC) every 8 weeks (Q8W) during Induction period.
- Induction: 30 mg Mirikizumab Q8W: Induction: Participants received 30 milligram (mg) mirikizumab SC Q8W during Induction period.
- Induction:100 mg Mirikizumab Q8W: Induction: Participants received 100 mg mirikizumab SC Q8W during Induction period.
- Induction: 300 mg Mirikizumab Q8W: Induction: Participants received 300 mg mirikizumab SC Q8W during Induction period.
- Maintenance: 30 mg Mirikizumab Q8W to 30 mg Mirikizumab PRN: Maintenance:
  Participants received 30 mg mirikizumab as needed (PRN) during the maintenance period.
  Participants who had greater than or equal to (≥) Psoriasis Area and Severity Index (PASI) 90 at Week 16 after receiving 30 mg mirikizumab Q8W during induction period.
  Follow-up: participants did not receive drug during the follow-up period.
- Maintenance: 100 mg Mirikizumab Q8W to 100 mg Mirikizumab PRN: Maintenance:
  Participants received 100 mg mirikizumab as needed (PRN) during the maintenance period.
  Participants had ≥ PASI 90 at Week 16 after receiving 100 mg mirikizumab Q8W during induction period.
  Follow-up: participants did not receive drug during the follow-up period.
- Maintenance: 300 mg Mirikizumab Q8W to 300 mg Mirikizumab PRN: Maintenance:
  Participants received 300 mg mirikizumab as needed (PRN) during the maintenance period.
  Participants had ≥ PASI 90 at Week 16 after receiving 300 mg mirikizumab Q8W during induction period.
  Follow-up: participants did not receive drug during the follow-up period.
- Maintenance: Placebo to 300 mg Mirikizumab Q8W: Maintenance:
  Participants received 300 mg mirikizumab Q8W during the maintenance period. Participants had received placebo during induction period.
  Follow-up: Participants did not receive drug during the follow-up period.
- Maintenance: 30 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W: Maintenance:
  Participants received 300 mg mirikizumab Q8W during the maintenance period. Participants had less than (<) PASI 90 at Week 16 after receiving 30 mg mirikizumab Q8W during induction period.
  Follow-up: Participants did not receive drug during the follow-up period.
- Maintenance: 100 mg Mirikizumab Q8W to 300 mg MirikizumabQ8W: Maintenance:
  Participants received 300 mg mirikizumab Q8W during the maintenance period. Participants had < PASI 90 at Week 16 after receiving 100 mg mirikizumab Q8W during induction period.
  Follow-up: participants did not receive drug during the follow-up period.
- Maintenance: 300 mg Mirikizumab Q8W: Maintenance:
  Participants who had < PASI 90 at Week 16 continued to receive 300 mg mirikizumab SC Q8W during maintenance period.
Period: Induction Period (16 Weeks)
Arm/Group | Induction: Placebo | Induction: 30 mg Mirikizumab Q8W | Induction:100 mg Mirikizumab Q8W | Induction: 300 mg Mirikizumab Q8W | Maintenance: 30 mg Mirikizumab Q8W to 30 mg Mirikizumab PRN | Maintenance: 100 mg Mirikizumab Q8W to 100 mg Mirikizumab PRN | Maintenance: 300 mg Mirikizumab Q8W to 300 mg Mirikizumab PRN | Maintenance: Placebo to 300 mg Mirikizumab Q8W | Maintenance: 30 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W | Maintenance: 100 mg Mirikizumab Q8W to 300 mg MirikizumabQ8W | Maintenance: 300 mg Mirikizumab Q8W
Started | 52 | 51 | 51 | 51 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 52 | 51 | 51 | 51 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 50 | 49 | 51 | 49 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Period (88 Weeks)
Arm/Group | Induction: Placebo | Induction: 30 mg Mirikizumab Q8W | Induction:100 mg Mirikizumab Q8W | Induction: 300 mg Mirikizumab Q8W | Maintenance: 30 mg Mirikizumab Q8W to 30 mg Mirikizumab PRN | Maintenance: 100 mg Mirikizumab Q8W to 100 mg Mirikizumab PRN | Maintenance: 300 mg Mirikizumab Q8W to 300 mg Mirikizumab PRN | Maintenance: Placebo to 300 mg Mirikizumab Q8W | Maintenance: 30 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W | Maintenance: 100 mg Mirikizumab Q8W to 300 mg MirikizumabQ8W | Maintenance: 300 mg Mirikizumab Q8W
Started | 0 (No participants received placebo during maintenance period.) | 0 (No participants received 30 mg mirikizumab Q8W in both induction and maintenance.) | 0 (No participants received 100 mg mirikizumab Q8W in both induction and maintenance.) | 0 | 15 (Participants received 30 mg mirikizumab Q8W during induction period.) | 30 (Participants received 100 mg mirikizumab Q8W during induction period.) | 34 (Participants received 300 mg mirikizumab Q8W during induction period.) | 50 (Participants received placebo during induction period.) | 34 (Participants received 30 mg mirikizumab Q8W during induction arm.) | 21 (Participants received 100 mg mirikizumab Q8W during induction arm.) | 15 (Participants received 300 mg mirikizumab Q8W during induction arm.)
Rescue Participants | 0 | 0 | 0 | 10 (In PRN not regaining ≥ PASI 90 after 3 consecutive doses of drug or have < PASI 50 after 1 dose.) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Roll Over to AMAH (NCT03556202) | 0 | 0 | 0 | 13 | 9 | 18 | 26 | 42 | 24 | 17 | 0
Completed | 0 | 0 | 0 | 0 | 13 | 27 | 30 | 45 | 30 | 19 | 13
Not Completed | 0 | 0 | 0 | 0 | 2 | 3 | 4 | 5 | 4 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 2 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 2 | 0 | 1
Period: Follow-Up (16 Weeks)
Arm/Group | Induction: Placebo | Induction: 30 mg Mirikizumab Q8W | Induction:100 mg Mirikizumab Q8W | Induction: 300 mg Mirikizumab Q8W | Maintenance: 30 mg Mirikizumab Q8W to 30 mg Mirikizumab PRN | Maintenance: 100 mg Mirikizumab Q8W to 100 mg Mirikizumab PRN | Maintenance: 300 mg Mirikizumab Q8W to 300 mg Mirikizumab PRN | Maintenance: Placebo to 300 mg Mirikizumab Q8W | Maintenance: 30 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W | Maintenance: 100 mg Mirikizumab Q8W to 300 mg MirikizumabQ8W | Maintenance: 300 mg Mirikizumab Q8W
Started | 0 | 0 | 0 | 0 | 2 (Not all participants that completed maintenance period continued to follow-up period.) | 4 (Not all participants that completed maintenance period continued to follow-up period.) | 3 (Not all participants that completed maintenance period continued to follow-up period.) | 3 (Not all participants that completed maintenance period continued to follow-up period.) | 6 (Not all participants that completed maintenance period continued to follow-up period.) | 2 (Not all participants that completed maintenance period continued to follow-up period.) | 0 (Not all participants that completed maintenance period continued to follow-up period.)
Completed | 0 | 0 | 0 | 0 | 2 | 4 | 3 | 3 | 6 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Induction: Placebo: Induction: Placebo administered SC Q8W during Induction period.
- Induction: 30 mg Mirikizumab: Induction: 30 mg Mirikizumab administered SC Q8W during Induction period.
- Induction: 100 mg Mirikizumab: Induction: 100 mg Mirikizumab administered SC Q8W during Induction period.
- Induction: 300 mg Mirikizumab: Induction: 300 mg Mirikizumab administered SC Q8W during Induction period.
- Total: Total of all reporting groups
Arm/Group | Induction: Placebo | Induction: 30 mg Mirikizumab | Induction: 100 mg Mirikizumab | Induction: 300 mg Mirikizumab | Total
Number analyzed (Participants) | 52 | 51 | 51 | 51 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (12.39) | 49.2 (13.28) | 46.0 (13.18) | 47.5 (13.23) | 47.2 (12.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 16 | 15 | 53
  Male | 42 | 39 | 35 | 36 | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 4 | 5 | 24
  Not Hispanic or Latino | 39 | 37 | 42 | 42 | 160
  Unknown or Not Reported | 5 | 7 | 5 | 4 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 7 | 7 | 6 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 3 | 3 | 8
  White | 44 | 43 | 41 | 42 | 170
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 4 | 7 | 7 | 5 | 23
  United States | 21 | 20 | 18 | 23 | 82
  Japan | 4 | 7 | 5 | 4 | 20
  Poland | 19 | 14 | 18 | 14 | 65
  Germany | 4 | 3 | 3 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥90% Improvement in Psoriasis Area and Severity Index (PASI 90)
Description: PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of scaling, redness, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no psoriasis (PsO) to 72 for the most severe disease. For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored separately and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs (0.4)]. Overall scores range from 0 (no PsO) to 72 (the most severe disease).
Time Frame: Week 16
Population: All participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction: Placebo | Induction: 30 mg Mirikizumab | Induction: 100 mg Mirikizumab | Induction: 300 mg Mirikizumab
Number analyzed (Participants) | 52 | 51 | 51 | 51
percentage of participants | 0 [0 to 0] | 29.4 [16.9 to 41.9] | 58.8 [45.3 to 72.3] | 66.7 [53.7 to 79.6]
Statistical Analysis 1: Comparison: Induction: Placebo vs Induction: 30 mg Mirikizumab; Test type: Superiority; p = 0.009, Regression, Logistic; Risk Difference (RD) = 29.4, 95% CI 2-sided [16.9 to 41.9]
Statistical Analysis 2: Comparison: Induction: Placebo vs Induction: 100 mg Mirikizumab; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 58.8, 95% CI 2-sided [45.3 to 72.3]
Statistical Analysis 3: Comparison: Induction: Placebo vs Induction: 300 mg Mirikizumab; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 66.7, 95% CI 2-sided [53.7 to 79.6]

2. Secondary Outcome: Percentage of Participants With a 100% Improvement in Psoriasis Area and Severity Index (PASI 100)
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of scaling, redness, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no PsO to 72 for the most severe disease. For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored separately and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor [head (0.1), upper limbs (0.2), trunk (0.3), lower limbs (0.4)]. Overall scores range from 0 (no PsO) to 72 (the most severe disease).
Time Frame: Week 16
Population: All participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction: Placebo | Induction: 30 mg Mirikizumab | Induction: 100 mg Mirikizumab | Induction: 300 mg Mirikizumab
Number analyzed (Participants) | 52 | 51 | 51 | 51
percentage of participants | 0 [0 to 0] | 15.7 [5.7 to 25.7] | 31.4 [18.6 to 44.1] | 31.4 [18.6 to 44.1]
Statistical Analysis 1: Comparison: Induction: Placebo vs Induction: 30 mg Mirikizumab; Test type: Superiority; p = 0.039, Regression, Logistic; Risk Difference (RD) = 15.7, 95% CI 2-sided [5.7 to 25.7]
Statistical Analysis 2: Comparison: Induction: Placebo vs Induction: 100 mg Mirikizumab; Test type: Superiority; p = 0.007, Regression, Logistic; Risk Difference (RD) = 31.4, 95% CI 2-sided [18.6 to 44.1]
Statistical Analysis 3: Comparison: Induction: Placebo vs Induction: 300 mg Mirikizumab; Test type: Superiority; p = 0.007, Regression, Logistic; Risk Difference (RD) = 31.4, 95% CI 2-sided [18.6 to 44.1]

3. Secondary Outcome: Percentage of Participants With a ≥75% Improvement in Psoriasis Area and Severity Index (PASI 75)
Description: as for outcome 2
Time Frame: Week 16
Population: All participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction: Placebo | Induction: 30 mg Mirikizumab | Induction: 100 mg Mirikizumab | Induction: 300 mg Mirikizumab
Number analyzed (Participants) | 52 | 51 | 51 | 51
percentage of participants | 3.8 [0 to 9.1] | 52.9 [39.2 to 66.6] | 78.4 [67.1 to 89.7] | 74.5 [62.5 to 86.5]
Statistical Analysis 1: Comparison: Induction: Placebo vs Induction: 30 mg Mirikizumab; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 22.49, 95% CI 2-sided [5.62 to 89.97]
Statistical Analysis 2: Comparison: Induction: Placebo vs Induction: 100 mg Mirikizumab; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 74.6, 95% CI 2-sided [62.1 to 87.0]
Statistical Analysis 3: Comparison: Induction: Placebo vs Induction: 300 mg Mirikizumab; Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 70.7, 95% CI 2-sided [57.6 to 83.7]

4. Secondary Outcome: Percentage of Participants With a Static Physician Global Assessment (sPGA) 0 and 0/1
Description: The sPGA is the physician's determination of the participant's PsO lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participant's PsO was assessed as 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe). An sPGA responder was defined as having a post-baseline sPGA score of "0" or "1" with at least a 2-point improvement from baseline. Participants who did not meet the clinical response criteria or had missing data at Week 16 were considered non-responders for non-responder Imputation (NRI) analysis.
Time Frame: Week 16
Population: All participants who received at least one dose of drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction: Placebo | Induction: 30 mg Mirikizumab | Induction: 100 mg Mirikizumab | Induction: 300 mg Mirikizumab
Number analyzed (Participants) | 52 | 51 | 51 | 51
percentage of participants
  sPGA (0) | 0 [0 to 0] | 15.7 [5.7 to 25.7] | 31.4 [18.6 to 44.1] | 31.4 [18.6 to 44.1]
  sPGA (0/1) | 1.9 [0 to 5.7] | 37.3 [24.0 to 50.5] | 70.6 [58.1 to 83.1] | 68.6 [55.9 to 81.4]
Statistical Analysis 1: Comparison: Induction: Placebo vs Induction: 30 mg Mirikizumab; sPGA (0); Test type: Superiority; p = 0.041, Regression, Logistic; Risk Difference (RD) = 15.7, 95% CI 2-sided [5.7 to 25.7]
Statistical Analysis 2: Comparison: Induction: Placebo vs Induction: 100 mg Mirikizumab; sPGA (0); Test type: Superiority; p = 0.007, Regression, Logistic; Risk Difference (RD) = 31.4, 95% CI 2-sided [18.6 to 44.1]
Statistical Analysis 3: Comparison: Induction: Placebo vs Induction: 300 mg Mirikizumab; sPGA (0); Test type: Superiority; p = 0.008, Regression, Logistic; Risk Difference (RD) = 31.4, 95% CI 2-sided [18.6 to 44.1]
Statistical Analysis 4: Comparison: Induction: Placebo vs Induction: 30 mg Mirikizumab; sPGA (0/1); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 35.3, 95% CI 2-sided [21.5 to 49.1]
Statistical Analysis 5: Comparison: Induction: Placebo vs Induction: 100 mg Mirikizumab; sPGA (0/1); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 68.7, 95% CI 2-sided [55.6 to 81.7]
Statistical Analysis 6: Comparison: Induction: Placebo vs Induction: 300 mg Mirikizumab; sPGA (0/1); Test type: Superiority; p < 0.001, Regression, Logistic; Risk Difference (RD) = 66.7, 95% CI 2-sided [53.4 to 80.0]

5. Secondary Outcome: Mean Change From Baseline on the Psoriasis Symptom Scale (PSS) Total Score
Description: PSS is a patient-administered assessment of 4 symptoms (itch, pain, stinging, and burning); 3 signs (redness, scaling, and cracking); and 1 item on the discomfort related to symptoms/signs. The overall severity for each individual symptom/sign from the patient's psoriasis is indicated by selecting the number from a numeric rating scale (NRS) of 0 to 10 that best describes the worst level of each symptom/sign in the past 24 hours, where 0=no symptom/sign and 10=worst imaginable symptom/sign. The total score was calculated by summing the 8 individual items and ranged from 0 to 80, higher scores indicated greater symptom/sign severity. Least Square(LS) Mean was calculated using Mixed Model Repeated Measures (MMRM) model with treatment, geographic region [United States/Outside United States (US/OUS)], previous therapy (yes/no), baseline value, visit, and the interaction treatment-by-visit as fixed factors, covariance structure = heterogeneous autoregressive.
Time Frame: Baseline, Week 16
Population: All participants who received at least one dose of study drug who had baseline and at least one post-baseline PSS observation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Induction: Placebo | Induction: 30 mg Mirikizumab | Induction: 100 mg Mirikizumab | Induction: 300 mg Mirikizumab
Number analyzed (Participants) | 43 | 43 | 44 | 44
units on a scale | -4.35 (2.29) | -31.19 (2.34) | -42.33 (2.37) | -33.66 (2.27)
Statistical Analysis 1: Comparison: Induction: Placebo vs Induction: 30 mg Mirikizumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -26.84, Standard Error of Mean 3.26
Statistical Analysis 2: Comparison: Induction: Placebo vs Induction: 100 mg Mirikizumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -37.99, Standard Error of Mean 3.29
Statistical Analysis 3: Comparison: Induction: Placebo vs Induction: 300 mg Mirikizumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -29.32, Standard Error of Mean 3.22

6. Secondary Outcome: Mean Change (Improvement) From Baseline on the Patient Global Assessment
Description: The Patient's Global Assessment of Disease Severity is a single-item participant-reported outcome measure on which participants are asked to rate the severity of their psoriasis "today" from 0 (Clear) = no psoriasis, to 5 (Severe) = the worst their psoriasis has ever been. Least Square (LS) Mean was calculated using Mixed Model Repeated Measures (MMRM) model with treatment, geographic region (US/OUS), previous therapy (yes/no), baseline value, visit, and the interaction treatment-by-visit as fixed factors, covariance structure = unstructured.
Time Frame: Baseline, Week 16
Population: All participants who received at least one dose of study drug who had baseline and at least one post-baseline Patient Global Assessment observation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Induction: Placebo | Induction: 30 mg Mirikizumab | Induction: 100 mg Mirikizumab | Induction: 300 mg Mirikizumab
Number analyzed (Participants) | 51 | 48 | 51 | 49
units on a scale | 0.35 (0.16) | 2.24 (0.16) | 2.91 (0.16) | 2.82 (0.16)
Statistical Analysis 1: Comparison: Induction: Placebo vs Induction: 30 mg Mirikizumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 1.90, Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Induction: Placebo vs Induction: 100 mg Mirikizumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 2.56, Standard Error of Mean 0.22
Statistical Analysis 3: Comparison: Induction: Placebo vs Induction: 300 mg Mirikizumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 2.47, Standard Error of Mean 0.22

7. Secondary Outcome: Mean Change From Baseline on the Dermatology Life Quality Index (DLQI) Total Score
Description: The DLQI is a patient-reported, 10-question, quality-of-life questionnaire that covers 6 domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include "Not at all," "A little," "A lot," and "Very much," with corresponding scores of 0, 1, 2, and 3 respectively. Questions 3-10 also have an additional response category of "Not relevant" which is scored as "0". For all questions, if unanswered the question is scored as "0". Totals range from 0 to 30 (less to more impairment). Least Square (LS) Mean was calculated using Mixed Model Repeated Measures (MMRM) model with treatment, geographic region (US/OUS), previous therapy (yes/no), baseline value, visit, and the interaction treatment-by-visit as fixed factors, covariance structure = unstructured.
Time Frame: Baseline, Week 16
Population: All participants who received at least one dose of study drug who had baseline and at least one post-baseline DLQI observation.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Induction: Placebo | Induction: 30 mg Mirikizumab | Induction: 100 mg Mirikizumab | Induction: 300 mg Mirikizumab
Number analyzed (Participants) | 51 | 48 | 51 | 49
score on a scale | -1.07 (0.69) | -9.19 (0.71) | -10.18 (0.69) | -9.64 (0.70)
Statistical Analysis 1: Comparison: Induction: Placebo vs Induction: 30 mg Mirikizumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -8.12, Standard Error of Mean 0.98
Statistical Analysis 2: Comparison: Induction: Placebo vs Induction: 100 mg Mirikizumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -9.11, Standard Error of Mean 0.97
Statistical Analysis 3: Comparison: Induction: Placebo vs Induction: 300 mg Mirikizumab; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -8.57, Standard Error of Mean 0.98

8. Secondary Outcome: Mean Change From Baseline on the 36-Item Short Form Health Survey (SF-36) Physical Component Summary (PCS) and Mental Component Summary (MCS) Scores
Description: The SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health, mental health, social functioning, vitality, and 2 component scores (MCS and PCS). MCS consisted of social functioning, vitality, mental health, and role-emotional scales. PCS consisted of physical functioning, bodily pain, role-physical, and general health scales. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with higher scores indicating better health status or functioning. Least Squares Mean (LS Mean) was calculated using Analysis of covariance (ANCOVA) model with treatment, geographic region (US/OUS), and previous therapy (yes/no) as fixed factors and baseline value as covariate.
Time Frame: Baseline, Week 16
Population: All participants who received at least one dose of study drug with a baseline value and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Induction: Placebo | Induction: 30 mg Mirikizumab | Induction: 100 mg Mirikizumab | Induction: 300 mg Mirikizumab
Number analyzed (Participants) | 51 | 48 | 51 | 49
score on a scale
  MCS | 0.28 (0.87) | 2.39 (0.90) | 2.74 (0.88) | 1.52 (0.88)
  PCS | 1.23 (0.84) | 4.58 (0.88) | 4.40 (0.85) | 5.09 (0.85)
Statistical Analysis 1: Comparison: Induction: Placebo vs Induction: 30 mg Mirikizumab; Mental Component Summary (MCS); Test type: Superiority; p = 0.009, ANCOVA; Mean Difference (Net) = 2.11, Standard Error of Mean 1.24
Statistical Analysis 2: Comparison: Induction: Placebo vs Induction: 100 mg Mirikizumab; Mental Component Summary (MCS); Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Net) = 2.74, Standard Error of Mean 1.22
Statistical Analysis 3: Comparison: Induction: Placebo vs Induction: 300 mg Mirikizumab; Mental Component Summary (MCS); Test type: Superiority; p = 0.087, ANCOVA; Mean Difference (Net) = 1.52, Standard Error of Mean 1.24
Statistical Analysis 4: Comparison: Induction: Placebo vs Induction: 30 mg Mirikizumab; Physical Component Summary; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 3.35, Standard Error of Mean 1.20
Statistical Analysis 5: Comparison: Induction: Placebo vs Induction: 100 mg Mirikizumab; Physical Component Summary; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 3.16, Standard Error of Mean 1.18
Statistical Analysis 6: Comparison: Induction: Placebo vs Induction: 300 mg Mirikizumab; Physical Component Summary; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 3.86, Standard Error of Mean 1.19

9. Secondary Outcome: Pharmacokinetics (PK): Area Under the Curve (AUC) of Mirikizumab From Baseline Through Week 104
Description: Pharmacokinetics (PK): Area Under the Curve (AUC) of Mirikizumab From Baseline through Week 104
Time Frame: Week 0, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 32, Week 40, Week 48, Week 52, Week 56, Week 64, Week 72, Week 80, Week 88, Week 96, Week 100, Week 104
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- 30 mg Mirikizumab Q8W to 30 mg Mirikizumab PRN: Participants received 30 mg mirikizumab as needed (PRN) during the maintenance period.
  Participants had ≥ PASI 90 at Week 16 after receiving 30 mg mirikizumab Q8W during induction period.
- 100 mg Mirikizumab Q8W to 100 mg Mirikizumab PRN: Participants received 100 mg mirikizumab as needed (PRN) during the maintenance period.
  Participants had ≥ PASI 90 at Week 16 after receiving 100 mg mirikizumab Q8W during induction period.
- 300 mg Mirikizumab Q8W to 300 mg Mirikizumab PRN: Participants received 300 mg mirikizumab as needed (PRN) during the maintenance period.
  Participants had ≥ PASI 90 at Week 16 after receiving 300 mg mirikizumab Q8W during induction period.
- Placebo to 300 mg Mirikizumab Q8W: Participants received 300 mg mirikizumab Q8W during the maintenance period.
  Participants had received placebo during induction period.
- 30 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W: Participants received 300 mg mirikizumab Q8W during the maintenance period.
  Participants had < PASI 90 at Week 16 after receiving 30 mg mirikizumab Q8W during induction period.
- 100 mg Mirikizumab Q8W to 300 mg MirikizumabQ8W: Participants received 300 mg mirikizumab Q8W during the maintenance period.
  Participants had < PASI 90 at Week 16 after receiving 100 mg mirikizumab Q8W during induction period.
- 300 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W: Participants received 300 mg mirikizumab SC Q8W during Induction period.
  Participants had < PASI 90 at Week 16 continued to receive 300 mg mirikizumab SC Q8W during maintenance period.
Arm/Group | 30 mg Mirikizumab Q8W to 30 mg Mirikizumab PRN | 100 mg Mirikizumab Q8W to 100 mg Mirikizumab PRN | 300 mg Mirikizumab Q8W to 300 mg Mirikizumab PRN | Placebo to 300 mg Mirikizumab Q8W | 30 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W | 100 mg Mirikizumab Q8W to 300 mg MirikizumabQ8W | 300 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W
Number analyzed (Participants) | 13 | 23 | 33 | 50 | 34 | 21 | 15
nanogram*hour per milliliter (ng*hr/mL) | 3.22 (46.33) | 8.94 (79.19) | 22.96 (55.80) | 46.4 (62.8) | 34.83 (92.13) | 47.66 (70.08) | 51.30 (43.54)

ADVERSE EVENTS:
Time Frame: Up To 120 Weeks
Description: All participants who received at least one dose of study drug.Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Induction: Placebo: Induction: Participants received placebo SC Q8W during Induction period.
- Induction: 30 mg Mirikizumab Q8W: Induction: Participants received 30 mg mirikizumab Q8W during Induction period.
- Maintenance: 30 mg Mirikizumab Q8W to 30 mg Mirikizumab PRN: Maintenance:
  Participants received 30 mg mirikizumab as needed (PRN) during the maintenance period.
  Participants who had ≥ PASI 90 at Week 16 after receiving 30 mg mirikizumab Q8W during induction period.
- Maintenance: 100 mg Mirikizumab Q8W to 100 mg Mirikizumab PRN: Maintenance:
  Participants received 100 mg mirikizumab as needed (PRN) during the maintenance period.
  Participants had ≥ PASI 90 at Week 16 after receiving 100 mg mirikizumab Q8W during induction period.
- Maintenance: 300 mg Mirikizumab Q8W to 300 mg Mirikizumab PRN: Maintenance:
  Participants received 300 mg mirikizumab as needed (PRN) during the maintenance period.
  Participants had ≥ PASI 90 at Week 16 after receiving 300 mg mirikizumab Q8W during induction period.
- Maintenance: Placebo to 300 mg Mirikizumab Q8W: Maintenance:
  Participants received 300 mg mirikizumab Q8W during the maintenance period. Participants had received placebo during induction period.
- Maintenance: 30 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W: Maintenance:
  Participants received 300 mg mirikizumab Q8W during the maintenance period. Participants had < PASI 90 at Week 16 after receiving 30 mg mirikizumab Q8W during induction period.
- Maintenance: 100 mg Mirikizumab Q8W to 300 mg MirikizumabQ8W: Maintenance:
  Participants received 300 mg mirikizumab Q8W during the maintenance period. Participants had < PASI 90 at Week 16 after receiving 100 mg mirikizumab Q8W during induction period.
- 300 mg Mirikizumab Q8W-Rescue: Participants received 300 mg Q8W mirikizumab during rescue.
- 30 mg Mirikizumab Q8W to 30 mg Mirikizumab PRN-Follow-up; 100 mg Mirikizumab Q8W to 100 mg Mirikizumab PRN-Follow-up; 300 mg Mirikizumab Q8W to 300 mg Mirikizumab PRN-Follow-up; Placebo to 300 mg Mirikizumab Q8W-Follow-up; 30 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W-Follow-up; 100 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W-Follow-up: Follow-up: Participants did not receive drug during the follow-up period.
Arm/Group | Induction: Placebo | Induction: 30 mg Mirikizumab Q8W | Induction:100 mg Mirikizumab Q8W | Induction: 300 mg Mirikizumab Q8W | Maintenance: 30 mg Mirikizumab Q8W to 30 mg Mirikizumab PRN | Maintenance: 100 mg Mirikizumab Q8W to 100 mg Mirikizumab PRN | Maintenance: 300 mg Mirikizumab Q8W to 300 mg Mirikizumab PRN | Maintenance: Placebo to 300 mg Mirikizumab Q8W | Maintenance: 30 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W | Maintenance: 100 mg Mirikizumab Q8W to 300 mg MirikizumabQ8W | Maintenance: 300 mg Mirikizumab Q8W | 300 mg Mirikizumab Q8W-Rescue | 30 mg Mirikizumab Q8W to 30 mg Mirikizumab PRN-Follow-up | 100 mg Mirikizumab Q8W to 100 mg Mirikizumab PRN-Follow-up | 300 mg Mirikizumab Q8W to 300 mg Mirikizumab PRN-Follow-up | Placebo to 300 mg Mirikizumab Q8W-Follow-up | 30 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W-Follow-up | 100 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W-Follow-up
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/51 | 0/51 | 0/51 | 0/15 | 0/30 | 0/34 | 0/50 | 0/34 | 0/21 | 0/15 | 0/10 | 0/2 | 0/4 | 0/3 | 0/3 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/52 | 1/51 | 0/51 | 1/51 | 1/15 | 2/30 | 1/34 | 2/50 | 2/34 | 2/21 | 3/15 | 1/10 | 0/2 | 0/4 | 0/3 | 0/3 | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 19/52 | 24/51 | 19/51 | 19/51 | 13/15 | 20/30 | 23/34 | 38/50 | 28/34 | 18/21 | 13/15 | 9/10 | 0/2 | 1/4 | 0/3 | 0/3 | 2/6 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction: Placebo (N=52) | Induction: 30 mg Mirikizumab Q8W (N=51) | Induction:100 mg Mirikizumab Q8W (N=51) | Induction: 300 mg Mirikizumab Q8W (N=51) | Maintenance: 30 mg Mirikizumab Q8W to 30 mg Mirikizumab PRN (N=15) | Maintenance: 100 mg Mirikizumab Q8W to 100 mg Mirikizumab PRN (N=30) | Maintenance: 300 mg Mirikizumab Q8W to 300 mg Mirikizumab PRN (N=34) | Maintenance: Placebo to 300 mg Mirikizumab Q8W (N=50) | Maintenance: 30 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W (N=34) | Maintenance: 100 mg Mirikizumab Q8W to 300 mg MirikizumabQ8W (N=21) | Maintenance: 300 mg Mirikizumab Q8W (N=15) | 300 mg Mirikizumab Q8W-Rescue (N=10) | 30 mg Mirikizumab Q8W to 30 mg Mirikizumab PRN-Follow-up (N=2) | 100 mg Mirikizumab Q8W to 100 mg Mirikizumab PRN-Follow-up (N=4) | 300 mg Mirikizumab Q8W to 300 mg Mirikizumab PRN-Follow-up (N=3) | Placebo to 300 mg Mirikizumab Q8W-Follow-up (N=3) | 30 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W-Follow-up (N=6) | 100 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W-Follow-up (N=2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enlarged uvula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal septal operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Induction: Placebo (N=52) | Induction: 30 mg Mirikizumab Q8W (N=51) | Induction:100 mg Mirikizumab Q8W (N=51) | Induction: 300 mg Mirikizumab Q8W (N=51) | Maintenance: 30 mg Mirikizumab Q8W to 30 mg Mirikizumab PRN (N=15) | Maintenance: 100 mg Mirikizumab Q8W to 100 mg Mirikizumab PRN (N=30) | Maintenance: 300 mg Mirikizumab Q8W to 300 mg Mirikizumab PRN (N=34) | Maintenance: Placebo to 300 mg Mirikizumab Q8W (N=50) | Maintenance: 30 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W (N=34) | Maintenance: 100 mg Mirikizumab Q8W to 300 mg MirikizumabQ8W (N=21) | Maintenance: 300 mg Mirikizumab Q8W (N=15) | 300 mg Mirikizumab Q8W-Rescue (N=10) | 30 mg Mirikizumab Q8W to 30 mg Mirikizumab PRN-Follow-up (N=2) | 100 mg Mirikizumab Q8W to 100 mg Mirikizumab PRN-Follow-up (N=4) | 300 mg Mirikizumab Q8W to 300 mg Mirikizumab PRN-Follow-up (N=3) | Placebo to 300 mg Mirikizumab Q8W-Follow-up (N=3) | 30 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W-Follow-up (N=6) | 100 mg Mirikizumab Q8W to 300 mg Mirikizumab Q8W-Follow-up (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (2) | 3 (15) | 3 (14) | 2 (9) | 1 (9) | 1 (6) | 1 (3) | 4 (92) | 3 (67) | 2 (31) | 0 (0) | 2 (39) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema migrans (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis a (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis e (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (8) | 5 (7) | 6 (8) | 8 (10) | 3 (8) | 3 (3) | 7 (10) | 15 (26) | 12 (25) | 5 (13) | 5 (12) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 6 (6) | 3 (3) | 2 (3) | 2 (2) | 5 (6) | 2 (2) | 8 (9) | 3 (7) | 5 (6) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethritis chlamydial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (5) | 1 (1) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0/10 (0) | 0/12 (0) | 0/16 (0) | 0/15 (0) | 0/4 (0) | 0/10 (0) | 1/8 (1) | 0/10 (0) | 0/8 (0) | 0/6 (0) | 0/6 (0) | 0/2 (0) | 0/0 (0) | 0/1 (0) | 0/1 (0) | 0/0 (0) | 0/3 (0) | 0/1 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0/10 (0) | 0/12 (0) | 0/16 (0) | 1/15 (1) | 0/4 (0) | 1/10 (1) | 0/8 (0) | 0/10 (0) | 0/8 (0) | 0/6 (0) | 0/6 (0) | 0/2 (0) | 0/0 (0) | 0/1 (0) | 0/1 (0) | 0/0 (0) | 0/3 (0) | 0/1 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (5) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (4) | 2 (2) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 8 (10) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (5) | 3 (3) | 3 (4) | 2 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/10 (0) | 0/12 (0) | 0/16 (0) | 0/15 (0) | 0/4 (0) | 0/10 (0) | 0/8 (0) | 0/10 (0) | 0/8 (0) | 0/6 (0) | 1/6 (1) | 0/2 (0) | 0/0 (0) | 0/1 (0) | 0/1 (0) | 0/0 (0) | 0/3 (0) | 0/1 (0)
Menorrhagia (Reproductive system and breast disorders) | 0/10 (0) | 0/12 (0) | 0/16 (0) | 0/15 (0) | 0/4 (0) | 0/10 (0) | 0/8 (0) | 1/10 (1) | 0/8 (0) | 0/6 (0) | 0/6 (0) | 0/2 (0) | 0/0 (0) | 0/1 (0) | 0/1 (0) | 0/0 (0) | 0/3 (0) | 0/1 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/10 (0) | 0/12 (0) | 0/16 (0) | 0/15 (0) | 0/4 (0) | 0/10 (0) | 0/8 (0) | 1/10 (1) | 0/8 (0) | 0/6 (0) | 0/6 (0) | 0/2 (0) | 0/0 (0) | 0/1 (0) | 0/1 (0) | 0/0 (0) | 0/3 (0) | 0/1 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0/42 (0) | 0/39 (0) | 0/35 (0) | 0/36 (0) | 0/11 (0) | 0/20 (0) | 0/26 (0) | 0/40 (0) | 0/26 (0) | 0/15 (0) | 1/9 (1) | 0/8 (0) | 0 (0) | 0/3 (0) | 0/2 (0) | 0 (0) | 0/3 (0) | 0/1 (0)
Scrotal pain (Reproductive system and breast disorders) | 0/42 (0) | 0/39 (0) | 0/35 (0) | 0/36 (0) | 0/11 (0) | 0/20 (0) | 0/26 (0) | 0/40 (0) | 0/26 (0) | 1/15 (1) | 0/9 (0) | 0/8 (0) | 0 (0) | 0/3 (0) | 0/2 (0) | 0 (0) | 0/3 (0) | 0/1 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/10 (0) | 0/12 (0) | 0/16 (0) | 0/15 (0) | 0/4 (0) | 1/10 (1) | 0/8 (0) | 0/10 (0) | 0/8 (0) | 0/6 (0) | 0/6 (0) | 0/2 (0) | 0/0 (0) | 0/1 (0) | 0/1 (0) | 0/0 (0) | 0/3 (0) | 0/1 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/10 (0) | 0/12 (0) | 0/16 (0) | 1/15 (1) | 0/4 (0) | 0/10 (0) | 0/8 (0) | 0/10 (0) | 0/8 (0) | 0/6 (0) | 0/6 (0) | 0/2 (0) | 0/0 (0) | 0/1 (0) | 0/1 (0) | 0/0 (0) | 0/3 (0) | 0/1 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 5 (8) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 3 (3) | 3 (4) | 4 (4) | 3 (3) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/88/NCT02899988/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT02899988/SAP_001.pdf